CLINICAL TRIAL: NCT06880497
Title: Monocentric, Randomized Study, Comparing Articular Noise and Its Perception Between Two Different Types of Total Knee Arthroplasty
Brief Title: Comparing Articular Noise and Its Perception Between Two Different Types of Total Knee Arthroplasty
Acronym: NATKA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-02452-45
Record Dates: First submitted 2025-03-04; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthristis; Knee Replacement Arthroplasty; Knee Replacement, Total
Keywords: Noise; Articular noise; Total Knee Arthroplasty; TKA; Total Knee Replacement; TKR
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Intervention Model Description: Prospective, monocentric, comparative, 1:1 randomized, single-blinded study evaluating the prevalence of articular noise following primary TKA using UC versus PS implants.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- UC TKA (Active Comparator): The Score II® is a primary cruciate-sacrificing TKA, with a single-radius femoral component that articulates in an ultra-congruent (UC) mobile-bearing tibial insert. The mobile-bearing tibial insert has high anterior and posterior borders to avoid anterior subluxation of the femoral condyles during knee flexion and a concave articular surface with a radius of curvature that matches that of the femoral component in the sagittal plane to ensure high congruence. The Score II® UC TKA comprises eight sizes and offers the choice of using a cemented or uncemented version. In this study, only the cemented version will be used.
  Interventions: Procedure: total knee arthroplasty
- PS TKA (Active Comparator): The Anatomic® is a primary PS TKA with a fixed-bearing polyethylene insert. The femoral component has a cam design that engages on a tibial post to provide anterior-posterior stability during flexion. The Anatomic® PS TKA comprises nine cemented sizes. In this study, only the cemented version will be used. The Anatomic® PS TKA comprises nine cemented sizes.
  Interventions: Procedure: total knee arthroplasty

INTERVENTIONS:
Procedure: total knee arthroplasty — Replacement of knee articulating surface for patients with end-stage osteoarthritis.
  Other Names: knee surgery; knee replacement

SUMMARY:
Some patients complain of articular noise (such as clicking, snapping, cracking or popping) after a total knee replacement. Controversy remains about whether there is a correlation between articular noise and worse outcomes following a knee replacement. A study by Nam et al. on 1540 patients revealed an association between noise and residual symptoms 30 days after they received a total knee replacement. Conversely, a study by Kuriyama et al. on 60 patients revealed no correlation between noise and patient satisfaction after 1 year of receiving a total knee replacement. The incidence of noise following a knee replacement has rarely been studied as a primary outcome. Like pain, it could be considered an important patient-reported outcome to assess patient satisfaction. The study aims to compare the prevalence of patient-perceived noise of an ultra-congruent total knee prosthesis (Score 2, Amplitude) versus a posterior-stabilized total knee prosthesis (Anatomic, Amplitude).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients receiving a primary TKA
* Signed informed consent
* Patients affiliated to a social security scheme
* Patients willing and able to comply with study protocol requirements based on the investigator's judgment.

Exclusion Criteria:

* History of knee surgery on the concerned/studied knee (except arthroscopic surgery)
* Patients presenting coronal deformities > 20°, varus laxity > 10° and/or valgus laxity > 15°
* Patients receiving revision TKA
* Pregnancy or breast-feeding
* Patients with protected status under articles L1121-6, LL121-8 and L1122-2 of the French Public Health Code
* Unable to comply with study procedures, based on the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of articular noise | 2 years
  The primary outcome is the prevalence of patients with articular noise at 2 years, evaluated by the Investigator during the follow-up visit through clinical examination and using the following question (Q1):
  Q1: Do you hear noise? Never, rarely, sometimes, often, extremely often

SECONDARY OUTCOMES:
Noise characterisation: Discomfort | 1 year and 2 years
  Characterisation of discomfort due to noise
  Q2: Do you feel noise? (Never, rarely, sometimes, often, extremely often) Q3: Is the noise a concern, causing discomfort? (Never, rarely, sometimes, often, extremely often)
Noise characterisation: Type | 1 and 2 years
  Characterisation of the type of noise:
  Q4: What kind of noise do you hear of feel? (Clunk, crepitus, grinding, clicking, other)
Noise characterisation: Location | 1 and 2 years
  Characterisation of the location of noise:
  Q5: What part of the knee is involved? (Patella, joint, both, other)
Noise characterisation: impact on quality of life | 1 and 2 years
  Characterisation of impact on quality of life:
  Q6: What is the impact of the noise on your quality of life, on a scale from 0 (none) to 10 (severe)?
Patient reported outcome score | 1 and 2 years
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC): worst, 96; best, 0

OTHER OUTCOMES:
Forgotten joint | 1 and 2 years
  Forgotten Joint Score (FJS): worst, 0; best, 100
Patient reported outcome score | 1 and 2 years
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC): worst, 96; best, 0
Knee mobility: Maximum flexion | 3 weeks, 3 months, 1 years and 2 years
  Clinical evaluation of knee mobility, using measurements of maximum flexion: degrees
Knee mobility: flexion contracture | 3 weeks, 3 months, 1 years and 2 years
  Clinical evaluation of knee mobility, using measurements of flexion contracture (FC): degrees
Knee mobility: Range of motion | 3 weeks, 3 months, 1 years and 2 years
  Clinical evaluation of knee mobility, using measurements of range of motion (ROM): degrees
Joint pain | 3 weeks, 3 months, 1 year and 2 years
  Pain assessment using the numeric scale (0 to 10): 0, no pain; 10, excruciating pain.
Patient satisfaction | 1 and 2 years
  Patient satisfaction assessed using a 5-point Likert scale (very satisfied, satisfied, neutral, dissatisfied, very dissatisfied).
Patient quality of life | 1 and 2 years
  Patient QoL using the EQ-5D-5L questionnaire: 0, worst; 1, best.
Adverse events | 0 to 2 years
  Analysis of adverse events: incidence, severity, and relationship to the medical device.

IPD SHARING:
Plan to Share IPD: Undecided
Upon a reasonable request, the authors will consider sharing anonymised data while adhering to French and European laws.

REFERENCES:
- [Background] Taniguchi H, Itoh M, Yoshimoto N, Itou J, Kuwashima U, Okazaki K. Noise after total knee arthroplasty has limited effect on joint awareness and patient-reported clinical outcomes: retrospective study. BMC Musculoskelet Disord. 2020 Feb 21;21(1):115. doi: 10.1186/s12891-020-3134-7. PMID 32085760
- [Background] Nam D, Barrack T, Nunley RM, Barrack RL. What Is the Frequency of Noise Generation in Modern Knee Arthroplasty and Is It Associated With Residual Symptoms? Clin Orthop Relat Res. 2017 Jan;475(1):83-90. doi: 10.1007/s11999-016-4701-y. PMID 26762299